CLINICAL TRIAL: NCT05685290
Title: The Effect of Pushing Technique With Saline on Success of Peripheral Intravenous Catheter Placement: A Randomized Controlled Study in a Pediatric Hematology and Oncology Sample
Brief Title: The Effect of Pushing Technique With Saline on Success of Peripheral Intravenous Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Meltem Gürcan, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 273
Record Dates: First submitted 2023-01-03; First posted 2023-01-17 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Nurse's Role
Keywords: Pediatric oncology; Intravenous Catheter Placement; nursing; randomized controlled study

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Participants will be blinded to group allocation and randomization process. Additionally they will be blinded for interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pushing with saline technique
  Interventions: Other: Pushing with saline technique
- Control group (Active Comparator): Traditional method
  Interventions: Other: Traditional method

INTERVENTIONS:
Other: Pushing with saline technique — Peripheral venous catheter placement by pushing with saline technique
  Arms: Intervention group
Other: Traditional method — Peripheral venous catheter placement with the traditional method by nurses in the clinic routinely.
  Arms: Control group

SUMMARY:
The aim of this project is to determine the effect of pushing with saline technique on the success of peripheral IV catheter placement in a pediatric hematology and oncology sample. This research is a randomized controlled experimental study.

DETAILED DESCRIPTION:
The sample of the study consists of children who aged 0-17. It is planned to collect the research data in Akdeniz University Hospital Pediatric Hematology and Oncology Outpatient Clinic. Data Collection Tools are 'Personal Information Form for Children', 'Catheterization Description Form' and 'The Difficult Intravenous Access (DIVA) Score for children '. DIVA Score will be used pre-intervention to determine whether patients have a difficult vein. Children with DIVA score of 4 and above will be randomly assigned to the intervention and control groups. The attempt to place an IV catheter in children in the intervention group will be carried out by "pushing with saline" (SF) technique. In this way, it is predicted that the success of IV intervention in difficult vascular access will increase and the number of attempts will decrease significantly. Peripheral catheter placement in the control group will be performed with the traditional method routinely implemented by nurses.

ELIGIBILITY:
Inclusion Criteria:

* The child who ages of 0-17.
* The child's need for peripheral IV catheter placement for treatment.
* A score of 4 or higher on the Difficult Intravenous Access Score for Children

Exclusion Criteria:

* None.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Catheterization Description Form | Immediately after the procedure.
  The form contains the catheter information regarding the children. It includes 7 questions including the time elapsed since the last vascular access, causes of catheter removal complications (infiltration, vascular damage, etc.), IV catheter location, IV catheter size (number), and peripheral vein where the catheter was placed. Primary endpoint of the study is Catheterization Description Form.

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan ATAY TURAN, PhD, Study Director — Assistant Professor; Ayla KAYA, PhD, Study Director — Research Assistant; Elif GÜLER, PhD, Study Director — Professor
Locations (1):
- Meltem Gürcan, Konyaalti, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurcan M, Karatas N, Kaya A, Turan SA, Guler E. The effect of a pushing technique with normal saline on peripheral intravenous catheter placement success in paediatric haematology and oncology: A randomized controlled trial. Eur J Oncol Nurs. 2024 Aug;71:102656. doi: 10.1016/j.ejon.2024.102656. Epub 2024 Jul 2. PMID 39002409